CLINICAL TRIAL: NCT05531760
Title: Predictive Factors of Graft Detachment Following Dmek: Retrospective Study About 170 Cases
Brief Title: Predictive Factors of Graft Detachment Following Dmek
Acronym: PDF DMEKDETACH
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-10Obs-CHRMT
Record Dates: First submitted 2022-09-02; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Fuchs' Endothelial Corneal Dystrophy; Descemet Membrane Endothelial Keratoplasty; Pseudophakic Bullous Keratopathy; Graft Detachment
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DMEK-operated eyes without graft detachment: Eyes operated with DMEK without graft detachment
  Interventions: Procedure: Descemet Membrane Endothelial Keratoplasty
- DMEK-operated with graft detachment: Eyes operated with DMEK with graft detachment
  Interventions: Procedure: Descemet Membrane Endothelial Keratoplasty

INTERVENTIONS:
Procedure: Descemet Membrane Endothelial Keratoplasty — DMEK-operated eyes

SUMMARY:
The aim of this study was to identify the predictive factors of graft detachment after Descemet Membrane Endothelial Keratoplasty (DMEK) surgery. This retrospective study was conducted on patients aged 18 years, with Fuchs' dystrophy (FECD) or pseudophakic bullous keratopathy (PBK), who were scheduled for DMEK or triple-DMEK (combined phacoemulsification and DMEK surgery). Patients with a history of surgery other than cataract surgery were excluded. The study was conducted between 2014 and 2022 and follow-up was for 3 months. The characteristics of patients with and without graft detachment following surgery were compared using logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with DMEK surgery

Exclusion Criteria:

* all associated eye surgery other than cataract surgery
* all existing anterior segment anomalies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with fuchs endothelial corneal dystrophy and patients with pseudophakic bullous keratopathies requiring corneal transplantation
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Appearence of the graft on anterior segment optical coherence tomography (AS OCT) examination | up to 3 months after surgery
  clinical examination and anterior segment optical coherence tomography (AS OCT) examination (appearence of the graft)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc PERONE, MD, Principal Investigator — CHR Metz Thionville Hopital de Mercy
Locations (1):
- CHR Metz-Thionville/Hopital de Mercy, Metz, France